CLINICAL TRIAL: NCT06540651
Title: Proof-of-concept Study on the Efficacy of Light Therapy in the Prophylactic Treatment of Chronic Cluster Headache
Brief Title: Efficacy of Light Therapy in Treatment of Chronic Cluster Headache
Acronym: LUMIAVFc
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RCAPHM23_0463; 2024-A01453-44 (Other: ID-RCB)
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-02

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group (group 1) (Experimental): Luminette® with active light emission in the 400 < X < 750 nm spectrum
  Interventions: Other: use of Luminettes ® with active light emission
- Control group (group 2) (Placebo Comparator): Luminette ® with modified spectral parameters for wavelengths covered, with light emission in a spectrum of 560 < X < 650 nm assumed to have no therapeutic effect (placebo effect)
  Interventions: Other: use of Luminettes ® with a light emission presumed to have no therapeutic effect

INTERVENTIONS:
Other: use of Luminettes ® with active light emission — Spectrum of 400 < X < 750 nm assumed active
  Arms: Experimental group (group 1)
Other: use of Luminettes ® with a light emission presumed to have no therapeutic effect — Modification of spectrum parameters for wavelengths covered, with light emission in a spectrum of 560 < X < 650 nm assumed to have no therapeutic effect
  Arms: Control group (group 2)

SUMMARY:
Cluster headache is a primary headache. The chronic form of the disease is often difficult to treat. It is now considered a chronobiological disease. This chronobiological character is based on clinical, biological and radiological arguments.

This study focuses on the use of light therapy in cluster headache. Light therapy has already been used in the treatment of other chronobiological diseases, such as seasonal depression, but also recently in the therapy of other primary headaches (such as migraine). Its aim is to re-adjust chronobiological rhythms, and it therefore seems worth testing in the chronic form of cluster headache.

Light therapy is delivered to the patient using a consumer electronics device.The main objective is to evaluate the prophylactic efficacy of light therapy in patients with chronic cluster headache.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of 18 years years old or more;
* Diagnosis of chronic cluster headache according to ICHD-3 criteria;
* Number of seizures during baseline equal to at least 24;
* Stability of prophylactic treatment for at least 1 month and commitment not to change it for the duration of the study;
* Patient affiliated to the French social security system.
* Patient who understands and speaks French correctly;
* Patient who has given free and informed written consent.

Exclusion Criteria:

* Contraindication to the use of light therapy: use of a photosensitizing treatment;
* Ophthalmological history: cataract, macular degeneration, glaucoma, retinitis pigmentosa;
* Patients who work at night;
* Other neurological, psychiatric or developmental pathologies considered incompatible with the study;
* Background treatment of cluster headache with melatonin;
* Persons protected by articles L1121-5, L1121-6 and L1121-8 of the French Public Health Code (pregnant or breast-feeding women, persons deprived of their liberty by judicial decision, socially vulnerable persons, adults incapable or unable to express their consent).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2027-02-05 (Estimated); Study Completion 2027-05-05 (Estimated)

PRIMARY OUTCOMES:
The median weekly number of cluster headache attacks | At day 28
  The difference in the median weekly number of cluster headache attacks between the month prior to randomization and the month of the double-blind period, between the two arms.

SECONDARY OUTCOMES:
Incidence and nature of adverse reactions | Daily
  Headache, eye fatigue, dry eyes, nausea
Intensity of cluster headache | Daily
  mild, moderate, severe, very severe
Use of acute treatments | Daily
  sumatriptan and oxygen therapy
Patient's Global Impression of Change (PGIC) score | At day 28
  From better outcome, score 1 (Highly improved) to worse outcome, score 7 (Highly aggravated)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital La Timone, Marseille
  - Hôpital de Cimiez, Nice

IPD SHARING:
Plan to Share IPD: No